CLINICAL TRIAL: NCT02361242
Title: 24-week Open-label Extension Study Evaluating the Effect of PXT00864 in Mild Alzheimer's Disease Patients Further to PLEODIAL-I Completion
Brief Title: 24-week Open-label Extension Study Evaluating PXT00864 Effect in Mild AD Patients Further to PLEODIAL-I Completion
Acronym: PLEODIAL-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharnext S.C.A. (Other)
Collaborators: Ascopharm Groupe Novasco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PXT00864-04
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2014-12

CONDITIONS: Alzheimer Disease
Keywords: PXT00864; mild AD; phase 2a
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PXT00864 Dose 1 (Experimental): 1 orange capsule containing 0.4 mg of acamprosate and 1 white capsule containing 6 mg of baclofen are taken orally b.i.d during 24 weeks.
  Interventions: Drug: PXT00864
- PXT00864 Dose 2 (Experimental): 1 orange capsule containing 1 mg of acamprosate and 1 white capsule containing 15 mg of baclofen are taken orally b.i.d during 24 weeks.
  Interventions: Drug: PXT00864
- PXT00864 Dose 3 (Experimental): 1 orange capsule containing 20 mg of acamprosate and 1 white capsule containing 12 mg of baclofen are taken orally b.i.d during 24 weeks.
  Interventions: Drug: PXT00864

INTERVENTIONS:
Drug: PXT00864 — PXT00864 is a fixed-dose combination of baclofen and acamprosate

SUMMARY:
PLEODIAL-II study is an extension of the previous pilot PLEODIAL-I study (CLN-PXT00864-03 protocol) and is designed for the descriptive analysis of patients with mild AD who are exposed to PXT00864 over an additional 24-week period.

DETAILED DESCRIPTION:
Patients having completed the previous 12-week PLEODIAL-I study were eligible to receive PXT00864 in this 24-week open-label extension PLEODIAL-II study in order to collect some additional long-term data regarding the safety and the potential effect of PXT00864 on cognitive and behavioural impairments.

ELIGIBILITY:
Main Inclusion Criteria:

* Mild Alzheimer's Disease patient who was included in PLEODIAL-I study
* Mini Mental State Examination (MMSE) score greater or equal to 20

Main Exclusion Criteria:

* Patient who was not compliant with the previous PLEODIAL-I study protocol
* Patient who experienced significant adverse events which necessitated treatment discontinuation during the PLEODIAL-I study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the total score of the 11-items Alzheimer's Disease Assessment Scale- Cognitive Subscale (ADAS-Cog) | V5 (study entry), V6 (after 12 weeks), V7 (after 24 weeks)
  Scores on the ADAS-Cog range from 0 to 70 with higher scores indicating greater cognitive impairment
Number of Treatment Emergent Adverse Events (TEAEs) | throughout the 24-week study period

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Orgogozo, MD, Principal Investigator — Hospital Pellegrin, Bordeaux, France
Locations (1):
- CMRR, Bordeaux, France, France